CLINICAL TRIAL: NCT07058974
Title: A Phase 1b, Multi-cohort Clinical Trial Assessing Safety and Feasibility of Exercise and Spermidine Administered in Conjunction With Lamivudine (RTi) or Rapamycin (mTORi) to Assess Impact on Dynamic Changes of Inflammation and Aging
Brief Title: A Study of Exercise and Pharmacologic Intervention on Systemic Inflammation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Thomas Marron, Director, Early Phase Trials Unit, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-24-01678
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Smokers; Former Smokers
MeSH Terms: conditions — Smoking Cessation | interventions — Lamivudine; Sirolimus; Spermidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise and spermidine administered in conjunction with lamivudine (RTi) (Experimental): Participants will perform an exercise regimen and take spermidine and lamivudine for 180 days.
  Interventions: Drug: lamivudine; Behavioral: Exercise Regimen; Dietary Supplement: Spermidine
- Exercise and spermidine administered in conjunction with rapamycin (mTORi) (Experimental): Participants will perform an exercise regimen and take spermidine and rapamycin for 180 days.
  Interventions: Drug: rapamycin; Behavioral: Exercise Regimen; Dietary Supplement: Spermidine

INTERVENTIONS:
Drug: lamivudine — Lamivudine (Epivir) is a drug used typically to treat HIV and Hepatitis B Virus (HBV). It has not been studied when given in combination with spermidine.
  Other Names: Epivir
  Arms: Exercise and spermidine administered in conjunction with lamivudine (RTi)
Drug: rapamycin — Rapamycin (Rapamune, Sirolimus) is an FDA-approved drug and indicated for use as an immune modulator.
  Other Names: Rapamune, Sirolimus
  Arms: Exercise and spermidine administered in conjunction with rapamycin (mTORi)
Behavioral: Exercise Regimen — All experimental groups will receive an exercise regimen combining high-intensity interval training (HIIT) (targeting aerobic fitness) and resistance training (targeting strength and skeletal muscle mass preservation). The HIIT exercise component will consist of 2 sessions per week totaling 20 minutes per session. The resistance training component will consist of 3 sessions per week totaling 40 minutes per session.
Dietary Supplement: Spermidine — Spermidine is a polyamine that forms naturally in plants, animals, and microorganisms as a byproduct of protein breakdown. Participants will take an oral dosage of 2mg/day for 180 days.

SUMMARY:
This is a study assessing the feasibility of performing an anti-aging intervention which is a combination of an exercise regimen, spermidine supplementation, and either rapamycin or lamivudine.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65-80 years old
* Current or former smokers
* BMI 25-32
* No cancer requiring active therapy within the last 2 years
* No autoimmune disease requiring disease modifying agents
* No patients with CKD stage 3/4 or ESRD
* No class 3 or 4 heart failure

Exclusion Criteria:

* Patients may not have cancer requiring active therapy within the last 2 years
* Patients may not have autoimmune disease requiring disease modifying agents
* Patients may not be receiving immune modifying biologic therapies
* Patients may not have chronic kidney disease stage 3/4 or end stage renal disease
* Patients may not have a known history of metabolic dysfunction-associated steatohepatitis
* Patients may not have a known chronic viral infection such as HIV or active Hepatitis B or C, or a known history of genital HSV. Patients who have spontaneously or through treatment cleared hepatitis B or C are candidates for the trial. If Hepatitis B core ab is positive must document a negative PCR.
* Patients may not have class 3 or 4 heart failure, or have experienced a myocardial infarction or cerebrovascular event in the past 6 months
* Patients may not have uncontrolled diabetes mellitus
* Patients may not have a history of clinically significant interstitial lung disease (ILD).
* Patients may not have clinically significant active wound healing due to recent injury or surgery
* Patients may not have signs or symptoms of clinically significant acute infectious illness on screening laboratory testing or physical examination.
* Patients may not have evidence of active or latent tuberculosis
* Patients may not have nephrotic range proteinuria on screening labs
* Patients may not have received a live virus within one month of study initiation.
* Patients cannot have uncontrolled hypertension (persistent systolic >160; diastolic >100)
* Patients with an inherited primary immunodeficiency
* Patients may not have a history of, or current evidence of, clinically significant chronic liver disease
* Patients may not be receiving any chronic immunosuppressive therapy.
* Patients may not be receiving medications that could increase rapamycin blood concentrations, such as strong inhibitors and inducers of CYP3A4 and/or P-gp (ketoconazole, voriconazole, itraconazole, erythromycin, telithromycin, or clarithromycin; rifampin or rifabutin), bromocriptine, cimetidine, cisapride, clotrimazole, danazol, diltiazem, fluconazole, protease inhibitors, metoclopramide, nicardipine, troleandomycin, verapamil. Furthermore, these medications may not be used during the study if patient is assigned to the rapamycin cohort.
* Patients may not be receiving medications that could decrease rapamycin blood concentrations, such as: carbamazepine, phenobarbital, phenytoin, rifapentine, St. John's Wort. Furthermore, these medications may not be used during the study if patient is assigned to the rapamycin cohort.
* Patients may not be receiving medications known to cause angioedema with concomitant use of rapamycin, such as angiotensin-converting enzyme (ACE) inhibitors. Furthermore, these medications may not be used during the study if patient is assigned to the rapamycin cohort.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number and Type of Grade 3/4 Adverse Events per CTCAE Version 5.0 | at 180 days
  Number and Type of Grade 3/4 Adverse Events per CTCAE Version 5.0. Toxicity will be assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0. Any patient experiencing a Grade 3 or 4 adverse event must hold drug until toxicity returns to grade 0-1. The treating investigator may hold study drug for any duration if the patient is deemed to be experiencing a Grade 1-2 adverse event related to study drug.
Number of participants with ability to complete >80% of specified pharmacological intervention | at 180 days
  Feasibility of the trial is determined by participant documentation of taking at least 80% of the provided study drug on a regular basis, ability to complete >80% of specified pharmacological intervention.

SECONDARY OUTCOMES:
Neutrophil to lymphocyte ratio (NLR) | at 180 days
  Measure NLR from complete blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marron, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to thomas.marron@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be determined).